CLINICAL TRIAL: NCT03979521
Title: Questionnaire Survey on the Systematic Recording and Characterization of Quality of Life Limitations in Myasthenia Gravis
Brief Title: Burden of Disease in Myasthenia Gravis
Acronym: Mya-BoD
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: NeuroCure Clinical Research Center, Charite, Berlin (Other)
Responsible Party: Principal Investigator, Andreas Meisel, Prof. Dr. med., Charite University, Berlin, Germany
Other Study IDs: Mya-BoD
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Myasthenia Gravis
Keywords: Myasthenia Gravis; Quality of life; Burden of disease; Social support
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Questionnaire-based survey addressed to german patients with the chronic autoimmune muscle disease called myasthenia gravis regarding quality of life, socioeconomic impact, social support, course of disease, complications of therapy and psychological comorbidities.

DETAILED DESCRIPTION:
Background:

Myasthenia gravis is a rare, chronic, antibody-mediated autoimmune disease that results in muscular weakness. The patients suffer from symptoms such as visual disturbances (especially double vision), weakness in the arms and legs, chewing and swallowing disorders and respiratory disorders, as well as crisis-related worsening of ventilation. This is often accompanied by pronounced fatigue (physical) and mental fatigue (depression).

Despite drug therapies that are on one hand symptomatic improving muscle strength, and on the other hand modulating the immune system, as well as specific procedures and drugs used in crises (plasmapheresis, immunoglobins) or refractory patients, patients are often severely limited, affecting everyday activities of self-care, family, social and professional life, thus affecting the mood and quality of life of patients. There is a lack of data measuring quality of life adequately.

Aim:

The aim of the data collection is to record the quality of life of myasthenia patients. By clinical information on the disease (including symptoms, course and therapy) and recording the social and occupational situation, the data should be contextualized. The following hypotheses are to be confirmed:

Primary hypotheses

* Myasthenia gravis affects the quality of life of patients comparable to neurological diseases such as multiple sclerosis
* Patients are limited in their participation in their private and professional life
* The severity of the disease is associated with the quality of life. Secondary hypotheses
* Myasthenia is associated with income busses and other economic disadvantages of the night
* Quality of life in myasthenia patients is related to fatigue and depression
* Quality of life in myasthenia patients depends on different therapy methods
* Myasthenia gravis has an impact on family planning and care for children.

Methods:

In cooperation with the German Myasthenia Gravis Society, a questionnaire prepared by the Charité will be sent to its members with a request for completion and an anonymous return. Similar projects have already been implemented in the past (response rate> 30%). About 3,300 patients should be contacted.

The returned questionnaires are then statistically evaluated and presented as part of a publication. For the evaluation of the hypotheses suitable descriptive, univariate analysis methods are used. Furthermore, with sufficient case numbers, multivariate analyzes (e.g., logistic regression) are also planned.

The questionnaire contains general information and questions about:

* Education and employment
* Social situation
* Social Support
* Economic aspects
* Symptoms and severity, course, treatment of myasthenia
* Quality of life
* Fatigue and depression

ELIGIBILITY:
Inclusion Criteria:

* Patients with Myasthenia Gravis
* Age ≥18 years

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Myasthenia Gravis being member at the German myasthenia gravis socitey (Deutsche Myasthenie Gesellschaft)
Sampling Method: Probability Sample
Enrollment: 1680 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Questionnaire for self-completion by patients containing questions about general information, information on myasthenia, information socioeconomic situation | directly after inclusion in the study
Hospital Anxiety and Depression Scale (HADS) | directly after inclusion in the study
  Questionnaire for self-completion by patients to determine the levels of anxiety and depression
Mya Quality of Life 15 (Mya QoL15) | directly after inclusion in the study
  Questionnaire for self-completion by patients for use as a measure of health outcome
Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF36) | directly after inclusion in the study
  Questionnaire for self-completion by patients for patients health
Myasthenia gravis Activities of daily living (MG ADL) | directly after inclusion in the study
  Questionnaire for self-completion by patients to determine symptom severity and limitations in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Meisel, Prof. Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- NeuroCure Clinical Research Center (NCRC), Charité University, Berlin, Mitte, Germany

REFERENCES:
- [Result] Lehnerer S, Jacobi J, Schilling R, Grittner U, Marbin D, Gerischer L, Stascheit F, Krause M, Hoffmann S, Meisel A. Burden of disease in myasthenia gravis: taking the patient's perspective. J Neurol. 2022 Jun;269(6):3050-3063. doi: 10.1007/s00415-021-10891-1. Epub 2021 Nov 20. PMID 34800167
- [Derived] Lehnerer S, Stegherr R, Grittner U, Stein M, Gerischer L, Stascheit F, Herdick M, Doksani P, Meisel A, Hoffmann S. The burden of disease in seronegative myasthenia gravis: a patient-centered perspective. Front Immunol. 2025 Apr 8;16:1555075. doi: 10.3389/fimmu.2025.1555075. eCollection 2025. PMID 40264778
- [Derived] Lehnerer S, Herdick M, Mevius A, Grittner U, Gansel P, Joeres L, Biskup J, Meisel A. The economic burden of Myasthenia gravis from the patient s perspective and reflected in German claims data. Sci Rep. 2025 Feb 25;15(1):6687. doi: 10.1038/s41598-025-91372-7. PMID 39994434
- [Derived] Stein M, Grittner U, Stegherr R, Gerischer L, Stascheit F, Hoffmann S, Herdick M, Legg D, Marbin D, Meisel A, Lehnerer S. The burden of myasthenia gravis - highlighting the impact on family planning and the role of social support. Front Neurol. 2023 Dec 14;14:1307627. doi: 10.3389/fneur.2023.1307627. eCollection 2023. PMID 38162439